CLINICAL TRIAL: NCT03720678
Title: A Phase 1/1b Study to Evaluate the Safety and Tolerability of Immunotherapy Combinations in Participants With Gastrointestinal Malignancies
Brief Title: A Study to Evaluate Immunotherapy Combinations in Participants With Gastrointestinal Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arcus Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ARC-3 (AB928CSP0003)
Record Dates: First submitted 2018-10-24; First posted 2018-10-25 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: GastroEsophageal Cancer; Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: 3+3 dose escalation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Escalation (Experimental): Dose escalation is a 3+3 design, including a Dose Limiting Toxicity (DLT) evaluation period. The RDE of etrumadenant will be determined in this part with escalating doses of etrumadenant in combination with the standard mFOLFOX chemotherapy regimen in participants with gastroesophageal or colorectal cancer.
  Interventions: Drug: etrumadenant; Drug: mFOLFOX
- Dose Expansion-GE (Experimental): The RDE of etrumadenant will be determined from the dose escalation part. Etrumadenant will be given in combination with the standard mFOLFOX chemotherapy regimen in participants with gastroesophageal cancer
  Interventions: Drug: etrumadenant; Drug: mFOLFOX
- Dose Expansion-CRC (Experimental): The RDE of etrumadenant will be determined from the dose escalation part. Etrumadenant will be given in combination with the standard mFOLFOX chemotherapy regimen in participants with colorectal cancer
  Interventions: Drug: etrumadenant; Drug: mFOLFOX

INTERVENTIONS:
Drug: etrumadenant — Etrumadenant is an A2aR and A2bR antagonist.
  Other Names: AB928
Drug: mFOLFOX — Oxaliplatin, Leucovorin and 5-fluorouracil given as part of standard mFOLFOX chemotherapy regimen

SUMMARY:
This is a Phase 1/1b, open-label, dose-escalation, and dose-expansion study to evaluate the safety, tolerability, pharmacokinetic (PK), pharmacodynamic (PD), and clinical activity of etrumadenant (AB928) in combination with mFOLFOX in participants with advanced metastatic gastroesophageal Cancer (GEC) or colorectal cancer (CRC).

DETAILED DESCRIPTION:
In the dose escalation phase, escalating doses of etrumadenant in combination with mFOLFOX at standard doses will be assessed in participants with advanced metastatic GEC or CRC. Eligible participants will receive oral administration of etrumadenant as well as IV infusion of mFOLFOX. The recommended dose for expansion (RDE) of etrumadenant will be determined upon completion of the dose-escalation phase.

In the dose expansion phase, etrumadenant at the RDE in combination with mFOLFOX at standard doses may be assessed in participants with advanced metastatic GEC or CRC.

Overall duration of treatment will depend on how well the treatment is tolerated. Treatment may continue until unacceptable toxicity or progressive disease or other reasons specified in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants ≥ 18 years
* Histologically confirmed gastroesophageal cancer or colorectal cancer that is metastatic, advanced or recurrent with progression
* Participants for whom mFOLFOX is considered appropriate therapy
* Must have at least 1 measurable lesion per RECIST v1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
* Must have received standard of care, including potentially curative available therapies or interventions.
* Confirm that an archival tissue sample is available and ≤ 24 months old; if not, a new biopsy of a tumor lesion must be obtained.
* Adequate organ and marrow function
* Previously treated central nervous system metastases, meeting the following criteria:

  * No evidence of progression by magnetic resonance imaging for at least 4 weeks prior to first dose.
  * Neurologic symptoms returned to baseline.
  * No immunosuppressive doses of systemic corticosteroids for at least 2 weeks before investigational product administration.
  * No carcinomatous meningitis.

Exclusion Criteria:

* Use of any live vaccines against infectious diseases (eg, influenza, varicella) within 4 weeks (28 days) of initiation of investigational product.
* Underlying medical conditions that, in the Investigator's or Sponsor's opinion, will make the administration of investigational product hazardous (eg interstitial lung disease, active infections requiring antibiotics, recent hospitalization with unresolved symptoms) or obscure the interpretation of toxicity determination or AEs, or concurrent medical condition requiring the use of immunosuppressive medications or immunosuppressive doses of systemic or absorbable topical corticosteroids.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the pre-screening or screening visit through 30 days after the last dose of etrumadenant in combination with mFOLFOX.
* Any active autoimmune disease or a documented history of autoimmune disease or syndrome that required systemic treatment in past 2 years (ie, with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs), except for vitiligo or resolved childhood asthma/atopy.

  * Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment.
  * Participants with asthma who require intermittent use of bronchodilators, inhaled corticosteroids, or local corticosteroid injections will not be excluded from this study. Participants on chronic systemic corticosteroids will be excluded from the study.
* Prior malignancy active within the previous 2 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix, breast, or prostate.
* Prior chemotherapy, targeted small-molecule therapy, or radiation therapy within 4 weeks prior to Day 1 or has not recovered (ie, ≥ Grade 1 or baseline) from AEs due to a previously administered agent, except ≤ Grade 2 alopecia or ≤ Grade 2 neuropathy and other AEs ≤ Grade 2 considered not clinically significant by the Medical Monitor and Investigator.
* Use of other investigational drugs (drugs not marketed for any indication) within 28 days of investigational product administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-11-18 (Actual); Primary Completion 2021-01-27 (Actual); Study Completion 2021-06-25 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | From first dose date to 90 days after the last dose (Approximately 1 year)
Incidence of dose-limiting toxicities (DLTs) during dose escalation phase | From first dose date to 28 days after the first dose

SECONDARY OUTCOMES:
Plasma concentration of etrumadenant | Recorded at baseline (prior to first dose), during the first 4 cycles of treatment (2 months), at end of treatment and 30 days post end of treatment (i.e. in total approximately 3 months)
Percentage of participants with Objective Response as determined by Investigator according to RECIST v1.1 | From study enrolment until participation discontinuation, first occurrence of progressive disease, or death from any cause, whichever occurs first (approximately 3-5 years)
Percentage of participants with Disease Control (complete response, partial response, or stable disease) for > 6 months as determined by RECIST v1.1 | From study enrolment until disease progression or loss of clinical benefit (up to approximately 3-5 years)
Duration of Response as determined by the Investigator according to RECIST v1.1 | From the date of first occurrence of a documented objective response to first documentation of disease progression or death from any cause, whichever occurs first (up to approximately 3-5 years)
Progression Free Survival (PFS) as determined by the Investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | From start of treatment up to first occurrence of progressive disease or death from any cause, whichever occurs first (up to approximately 3-5 years)
Overall Survival (OS) as determined by the Investigator according to RECIST v1.1 | From start of treatment up to death from any cause (up to approximately 3-5 years)
Receptor Occupancy in peripheral blood | Cycle 1 Day 1 through Cycle 4 Day 1 (2 months), at end of treatment and 30 days after end of treatment (in total approximately 3 months). Each Cycle is 14 days.
Immunomodulatory activity in subsets for AB928 in combination with mFOLFOX | Cycle 1 Day 1 through Cycle 4 Day 1 (2 months), at end of treatment and 30 days after end of treatment (in total approximately 3 months). Each Cycle is 14 days.
  Immunomodulatory activity will be assessed by aggregating data from biomarkers collected from peripheral blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Arcus Biosciences, Inc.
Locations (24):
- United States (17):
  - Arizona Clinical Research Center, Tucson, Arizona
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Maryland Oncology Hematology, Rockville, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - QUEST Research Institute, Farmington Hills, Michigan
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Carolina BioOncology Institute, Huntersville, North Carolina
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Prisma Health, Greenville, South Carolina
  - Texas Oncology - Austin Midtown, Austin, Texas
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology - Fort Worth Cancer Center, Fort Worth, Texas
  - Texas Oncology - San Antonio Northeast, San Antonio, Texas
  - Texas Oncology - San Antonio Medical Center, San Antonio, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
- Australia (7):
  - Border Medical Oncology, Albury, New South Wales
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - The Kinghorn Cancer Centre, Darlinghurst, New South Wales
  - St. George Private Hospital, Kogarah, New South Wales
  - Macquarie University Hospital, Macquarie Park, New South Wales
  - Peninsula & South Eastern Haematology and Oncology Group, Frankston, Victoria
  - Cabrini Hospital, Malvern, Victoria

IPD SHARING:
Plan to Share IPD: Yes
Arcus will provide access to individual de-identified participant data and related study documents (e.g., protocol, Statistical Analysis Plan [SAP], Clinical Study Report [CSR]) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions.
  For more information, please visit our website.
Supporting Information: Study Protocol, SAP, CSR
URL: https://trials.arcusbio.com/our-transparency-policy

REFERENCES:
- See also: ARC-3 - Lay Summary (English Version) — https://trials.arcusbio.com/study/?id=ARC-3